CLINICAL TRIAL: NCT00384280
Title: An Open Label, 2-period, Sequential Study to Determine the Impact of Multiple Doses of Rifampin on Single-dose Pharmacokinetics of HCV-796
Brief Title: Study to Determine the Impact of Multiple Doses of Rifampin on Single-dose Pharmacokinetics of HCV-796
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3173A1-110
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
MeSH Terms: interventions — Rifampin

INTERVENTIONS:
Drug: Rifampin

SUMMARY:
An open label, 2-period, sequential study to determine the impact of multiple doses of rifampin on single-dose pharmacokinetics of HCV-796

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of multiple oral doses of rifampin on the pharmacokinetic (PK) profile of a single oral dose of HCV-796 in healthy subjects.

SECONDARY OUTCOMES:
To assess the safety and tolerability of HCV-796 and rifampin when coadministered to healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer